CLINICAL TRIAL: NCT02912273
Title: Optimizing Fall-risk Prediction in Older Adults With Cancer
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 201609049
Record Dates: First submitted 2016-09-21; First posted 2016-09-23 (Estimated); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Cancer
Keywords: Geriatric assessment
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Fall Risk Assessment Group: -Participants will complete baseline primarily self-administered cancer-specific geriatric assessments and measures of neuropathy and pain, an abbreviated geriatric assessment with each follow-up clinic visit (generally every 3-4 weeks in patients receiving systemic therapy) for 6-months of follow-up and a final end-of-study assessment.
  Interventions: Other: Baseline Participant Assessment; Other: Baseline Healthcare Provider Assessment; Other: Follow-up Participant Assessment; Other: Follow-up Healthcare Provider Assessment; Other: End-of-study Participant Assessment; Other: End-of-study Healthcare Provider Assessment

INTERVENTIONS:
Other: Baseline Participant Assessment — * Section 1 contains demographic questions
  * Section 2 contains daily activity questions with multiple choice answers, multiple physical function questions, and if the participants has fallen and how many falls have occurred in the last 6 months
  * Section 3 has the participant list all medication
  * Section 4 contains several questions about participant health (lists of illnesses and indicate if illness interferes with their activities)
  * Section 5 contains several questions about participant fall concerns with answers ranging from 1=Not at all to 4=Very
  * Section 6 contains multiple questions asking about emotional distress/depression, fatigue, pain interference, pain intensity, and numbness and tingling
Other: Baseline Healthcare Provider Assessment — * Cognition: Orientation-Memory-Concentration Test which contains 6 questions that the provider will ask the participant. Form items 1-3, the response is either correct (score 0) or incorrect (score 1). For items 4-6, subtract one point for each error. Total score of 11 or greater indicates cognitive impairment (maximum score =28)
  * Trail Making Test Part B - consists of 25 circles distributed over a sheet of paper. The circles include both numbers and letters; the participants draws lines to connect the circles in an ascending pattern, but with the added task of alternating between the numbers and letter. The test is timed.
  * Timed "Up and "Go - the provider measures the time in seconds it takes for the participant to stand up from a standard arm chair, walk a distance of 3 meters, turn, walk back to the chair, and sit down again.
Other: Follow-up Participant Assessment — * Section 1 contains multiple choice questions about daily actives and several physical function questions
  * Section 2 asks the participants how many medications they take on a daily basis, indicate any medication for depression, anxiety, nausea , and other stomach conditions
  * Section 3 contains multiple questions asking about emotional distress/depression, fatigue, pain interference, pain intensity, and numbness and tingling
Other: Follow-up Healthcare Provider Assessment — * Trail Making Test Part B - consists of 25 circles distributed over a sheet of paper. The circles include both numbers and letters; the participants draws lines to connect the circles in an ascending pattern, but with the added task of alternating between the numbers and letter. The test is timed.
  * Timed "Up and "Go - the provider measures the time in seconds it takes for the participant to stand up from a standard arm chair, walk a distance of 3 meters, turn, walk back to the chair, and sit down again.
Other: End-of-study Participant Assessment — * Section 1 contains multiple choice questions about daily actives and several physical function questions
  * Section 2 asks the participants how many medications they take on a daily basis, indicate any medication for depression, anxiety, nausea , and other stomach conditions
  * Section 3 contains multiple questions about the participant's concern about falling with answers ranging from 1=Not at all to 4=Very
  * Section 4 contains multiple questions asking about emotional distress/depression, fatigue, pain interference, pain intensity, and numbness and tingling
Other: End-of-study Healthcare Provider Assessment — * Cognition: Orientation-Memory-Concentration Test which contains 6 questions that the provider will ask the participant. Form items 1-3, the response is either correct (score 0) or incorrect (score 1). For items 4-6, subtract one point for each error. Total score of 11 or greater indicates cognitive impairment (maximum score =28)
  * Trail Making Test Part B - consists of 25 circles distributed over a sheet of paper. The circles include both numbers and letters; the participants draws lines to connect the circles in an ascending pattern, but with the added task of alternating between the numbers and letter. The test is timed.
  * Timed "Up and "Go - the provider measures the time in seconds it takes for the participant to stand up from a standard arm chair, walk a distance of 3 meters, turn, walk back to the chair, and sit down again.

SUMMARY:
To establish the optimal strategy of fall-risk assessment to predict falls in older adults receiving cancer therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥65
* Receiving systemic cancer therapy, including conventional chemotherapy, novel/targeted agents or hormonal agents (e.g. anti-estrogen or anti-androgen) OR will begin systemic therapy within the next 4 weeks.
* Estimated life expectancy >1 year
* Anticipated to receive ongoing care at Siteman Cancer Center and its satellite sites
* Able to understand and willing to sign an IRB-approved written informed consent document

Exclusion Criteria:

* Unable to read and understand English

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Older adults receiving systemic therapy at Siteman Cancer Center
Sampling Method: Non-Probability Sample
Enrollment: 227 (Actual)
Dates: Start 2016-10-12 (Actual); Primary Completion 2020-01-09 (Actual); Study Completion 2020-01-09 (Actual)

PRIMARY OUTCOMES:
Number of falls | Up to 6 months
  -The Prevention of Falls Network Europe (PROFANE) Consensus Group guidelines will be used

SECONDARY OUTCOMES:
Time to fall event | Up to 6 months
Overall survival | Up to 6 months
Number of falls that were considered injurious falls | Up to 6 months
Fear of falling as Measured by the Falls Efficacy Scale-International | Up to 6 months
  measures the level of concern about falling during social and physical activities inside and outside the home whether or not the person actually does the activity. The level of concern is measured on a four point Likert scale (1=not at all concerned to 4=very concerned)

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Clifton, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu